CLINICAL TRIAL: NCT06326034
Title: Impact of Dapagliflozin as Add-on Therapy on Glycemic Status and Quality of Life in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohammed Mahmood Mohammed (Other)
Responsible Party: Sponsor-Investigator, Mohammed Mahmood Mohammed, Mohammed Mahmood Mohammed, Al-Mustansiriyah University
Organization: Al-Mustansiriyah University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAA234
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Nephropathy Type 2
MeSH Terms: interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: This interventional randomized clinical study was conducted from May to December 2022, at the National Diabetic Centre for treatment and research/ Mustansiriyah University/ Baghdad/ Iraq. Ethical approval from the diabetic center and college of pharmacy/ Mustansiriyah University, was taken prior to the study initiation. All investigations/ procedures carried out in this study involving human participants were in accordance with the 1975 Declaration of Helsinki and its later amendments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin group (Experimental): The study's outcomes measured the changes pre- and post-treatment with Dapagliflozin (week 0 to weeks 16). The following parameters being measured: HbA1c, fasting plasma glucose (FPG), postprandial plasma glucose (PPG; glucose level measured 2 hours after standardized breakfast), body weight (BW), height (Ht), waist circumference (WC), body mass index (BMI), index of central obesity (ICO), and patients' QoL.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 5 mg orally given once daily for four months.

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a syndrome of metabolic dysregulation that needs a multifactorial behavioral and pharmacological treatments to prevent or delay complications, morbidity and mortality. Uncontrolled hyperglycemia can be negatively affecting the patient's physical and psychological status and thus lower the patient's quality of life (QoL) (Verma & Dadarwal, 2017)(Vanstone et al., 2015)(Gebremedhin et al., 2019). According to American Diabetes Association (ADA), when hyperglycaemia remain uncontrolled (HbA1c ≥1.5% above the glycemic target), a second therapy for T2DM is needed (Davies et al., 2022).

It has been certained by ADA, beside the glucose lowering effect the add-on antidibetic medication should have an impact on weight management to achieve and maintain the optimum glycemic and weight control which are the goals in people without established cardiorenal risks (Vijan et al., 2014((Inzucchi et al., 2012). Although metformin still the first-line pharmacotherapy in most T2DM patients, according to American Diabetes Association (ADA) (Association, 2020) but has little or even weight neutral effect, as well as gliptins (Hermansen & Mortensen, 2007)(Sazan et al., 2012). Other old antidibetic classes such as thiazolidinediones (TZDs) and sulfonylureas (SUs) inspite of their efficacy in controlling glycemia but their use is associated with weight gain and other adverse effects (Derosa & Maffioli, 2010)(Najim et al., 2014)(Fonseca, 2003). However, The newest class of antidibetic drugs, sodium-glucose cotransporter 2 inhibitors (SGLT2i), are approved for the treatment of T2DM as add-on or even initial therapy (Tamez-Pérez et al., 2013). This class is act by inducing glycosuria and thus improving glycemic status without affecting insulin level (Merovci et al., 2015). Dapagliflozin is a highly selective inhibitor of SGLT2. It has been well tolerated and its safety and efficacy approved in the clinical trials, mostly on cardio-renal outcomes with additional benefits of weight loss and low risk of hypoglycemia (Heerspink et al., 2020)(Solomon et al., 2022)(Wiviott et al., 2019)(McMurray et al., 2019). To date, no clinical data regarding SGLT2i recorded in Iraqi patients with limited data available on Arabic population. On Qatari, assessment of Dapagliflozin effectiveness revealed a significant improvement in the glycemic status after 6 months when used in combination with standard therapy, a reduction (Al AdAwi et al., 2019). In Saudi Arabia, Dapagliflozin was found to be well-tolerated and effective treatment option for T2DM patients after 6 months (Alguwaihes, 2021).

DETAILED DESCRIPTION:
This interventional randomized clinical study was conducted from May to December 2022, at the National Diabetic Centre for treatment and research/ Mustansiriyah University/ Baghdad/ Iraq. Ethical approval from the diabetic center and college of pharmacy/ Mustansiriyah University, was taken prior to the study initiation. All investigations/ procedures carried out in this study involving human participants were in accordance with the 1975 Declaration of Helsinki and its later amendments.

Participants Recruitment Patients enrolled in the study with the following criteria: T2DM patients, age between 18-70 years, on a combination of OADs (sulfonylurea + metformin + gliptin) for at least 8 weeks before enrolment. Patients involved had an elevated glycosylated hemoglobin A1c (HbA1c) [7%-12.0%] at the time of enrollment. Patients who met the inclusion criteria and agreed to the study protocol were recruited, a written consent was obtained from all participants before starting the study. All patients involved were received Dapagliflozin 5mg once daily for 16 weeks. Sulfonylurea could be down-titrated only once during the treatment period to mitigate the risk of recurrent hypoglycemic events at the discretion of the investigator. Initially, 45 participant who met the criteria involved in the study and finished all the baseline requirement. At the end of the study, five cases recruited and the most with the commonest reasons for discontinuation being non-adherent with the study medication (1 case), non-compliance with the appointment (2 cases) and adverse events (2 cases of genitourinary infection). A total of 40 patients were completed the study.

ELIGIBILITY:
Inclusion Criteria:

* elevated glycosylated hemoglobin A1c (HbA1c) [7%-12.0%] at the time of enrollment

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life Assessment tool | the QOLSID was administered to the participants at study initiation (week 0) and after 16 weeks of study initiation.
  The QOLSID tool, introduced in 2020 by Mikhael EM et al. (Mikhael et al., 2020), was used in this study to measure the QoL in T2DM. The questionnaire consisted of 10 questions with 5 likert scale answers ranging from (0-4). Scores more than 32.5 indicates a good quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed Mahmood Mahmood, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No